CLINICAL TRIAL: NCT05197946
Title: Anatomical and Functional Imaging Correlates of Chronic Pain in Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other); Mount Washington Pediatric Hospital (Unknown); Neurosurgery Pain Research Institute (Unknown); Cerebral Palsy Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00181801
Record Dates: First submitted 2021-12-14; First posted 2022-01-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy; Chronic Pain
MeSH Terms: conditions — Cerebral Palsy; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with CP (survey-only): Subjects in this group are age 8 and older with a diagnosis of cerebral palsy. Participants are either able to affirmatively consent or assent with LAR consent. This sample will have a CFCS score ranging between 1 and 3 and should be able to unambiguously respond to a 65 item multiple choice survey.
- Neurotypical participants (survey-only): Subjects in this group are age 8 and older with no clinically significant neurologic or developmental diagnosis. Participants are either able to affirmatively consent or assent with LAR consent.
- Participants with CP (Survey + MRI): Subjects are 8 years or older with a diagnosis of cerebral palsy and clinical imaging demonstrating isolated periventricular white matter injury. Clinical assessment states that neurologic symptoms are attributed to this isolated injury. Subjects in this group must be able to lie still in a scanner for 1.5 hours in at most 2 sessions and be able to have an MRI. Participants must be able to affirmatively consent or assent with LAR consent.
  Interventions: Diagnostic Test: MRI
- Neurotypical participants (Survey + MRI): Subjects in this group are age 8 and older with no clinically significant neurologic or developmental diagnosis. Participants are able to affirmatively consent and are able to have an MRI. Subjects also should be able to lie still in a scanner for 1.5 hours.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Research unsedated MRI scans (outside of usual care) will be performed using a 3T Philips scanner at the F.M. Kirby Research Center. An MRI scanning protocol will be at the F.M. Kirby Research Center; the protocol will not last more than 1.5 hours. Acquisitions will include a triplanar survey, functional and anatomical multi-slice imaging of the brain as well as MRI of selected spinal levels. Protocols will be used that do not involve use of contrast agents and limit power/tissue absorption as well as otherwise remain within FDA and Kirby Center safety regulations. When possible, MRI will be performed within 3 months of initial survey/interview administration. If MRI is scheduled >3 months after initial survey/interview administration, a brief survey will be re-administered to screen for changes in pain/clinical status.
  Groups: Neurotypical participants (Survey + MRI); Participants with CP (Survey + MRI)

SUMMARY:
The investigators hope to use MRI biomarkers to identify and characterize sensorimotor network disruption patterns associated with chronic pain and sensory deficits in CP. Investigators will use existing information in the medical record as well as subjective reports from interview, physical exam data, and anatomical and functional MRI data to non-invasively identify brain injury correlates of pain and sensory deficits.

DETAILED DESCRIPTION:
Background: Seventy percent of adults with cerebral palsy (CP) have chronic pain. Patterns in pain symptoms suggest that different individuals have different types of pain. People with CP have differences in brain structure and function, but links with pain mechanisms are not well-understood. Better understanding could help inform precision diagnosis and management of pain subtypes in individuals with CP.

Objectives:

Primary: Identify and characterize sensorimotor network disruption patterns associated with chronic pain and motor deficits in CP

Secondary:

* Improve understanding of anatomical brain network changes in CP associated with sensory deficits and pain
* Identify non-invasive imaging-based neurobiomarkers applicable to sensory loss and pain in CP

Procedures:

Standardized online questionnaires: Participants (individuals with CP, controls, and/or caregivers) are first asked to complete standardized questionnaires reviewing pain symptoms, demographics, and medical history (CP-related and more generally). Online questionnaires replaced Structured Interview and Physical Examination procedures at the onset of COVID safety restrictions.

Review of medical records: For consenting individuals, medical records will be requested and reviewed by the research team. Previously-acquired traditional MRI obtained for clinical purposes will be requested and reviewed to detect correlation between routine neuroimaging markers of perinatal brain injury and CP and pain. If of suitable quality, quantitative analysis methods (e.g. analysis of brain lobe and ventricular volumes for volumetric anatomical sequences, analysis of white matter volumes from DTI sequences) may be applied to prior images.

MRI: Research unsedated MRI scans (outside of usual care) will be performed using a 3T Philips scanner at the F.M. Kirby Research Center. An MRI scanning protocol will be at the F.M. Kirby Research Center; the protocol will not last more than 1.5 hours. Acquisitions will include a triplanar survey, functional and anatomical multi-slice imaging of the brain as well as MRI of selected spinal levels. Protocols will be used that do not involve use of contrast agents and limit power/tissue absorption as well as otherwise remain within FDA and Kirby Center safety regulations. When possible, MRI will be performed within 3 months of initial survey/interview administration. If MRI is scheduled >3 months after initial survey/interview administration, a brief survey will be re-administered to screen for changes in pain/clinical status.

ELIGIBILITY:
Participants with CP (Survey-only):

Inclusion Criteria:

* Individual 8+ years of age
* Diagnosis of cerebral palsy

Exclusion Criteria:

-None

Neurotypical participants: (Survey-only):

Inclusion Criteria:

* Individual 8+ years of age
* Adult subject able to indicate understanding and affirmative consent OR Adult/child subject unable to indicate understanding and affirmative consent AND subject assents AND LAR consents

Exclusion Criteria:

-Clinically-significant neurologic or developmental diagnosis

Participants with CP (Survey and MRI):

Inclusion Criteria:

* Individual 8+ years of age
* Adult subject able to indicate understanding and affirmative consent OR Adult subject unable to indicate understanding and affirmative consent AND subject assents AND LAR consents
* Diagnosis of cerebral palsy
* Clinical imaging demonstrating isolated periventricular white matter injury
* Clinical judgment that all neurologic symptoms are attributable to non-progressive periventricular white matter injury
* Able to lie still in scanner for 1.5 hours in at most 2 sessions and be able to have MRI

Exclusion Criteria:

-None

Neurotypical participants (Survey and MRI):

Inclusion Criteria:

* Individual 8+ years of age
* Adult subject able to indicate understanding and affirmative consent
* Able to lie still in scanner for 1.5 hours and be able to have MRI

Exclusion Criteria:

-Clinically-significant neurologic or developmental diagnosis

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with cerebral palsy and typically-developing adults and children
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Regional brain/spine volumes | <3 months
  Regional volumes will be measured using MR processing software
Diffusion scalars | <3 months
  Diffusion scalars for tracts of interest including the posterior thalamic radiations as well as somatosensory association fibers and the spinothalamic tract

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chin, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (4):
- United States (4):
  - F.M. Kirby Center, Baltimore, Maryland
  - Mt. Washington Pediatric Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05197946/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT05197946/ICF_001.pdf